CLINICAL TRIAL: NCT06428747
Title: Investigating Microparticle Levels In Filtered Packed Red Blood Cell Units
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doha Fahmy, Assistant lecturer, Assiut University
Other Study IDs: Doha Sholkamy
Record Dates: First submitted 2024-05-13; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Packed Red Cells Causing Adverse Effects in Therapeutic Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 30 filtered backed RBCs.: detection of micro-particles.
  Interventions: Diagnostic Test: b. Detection of micro particles and their subtypes by flow cytometery on(BECKMAN COULTER CytoFLEX flow cytometer).
- 30 non-filtered backed RBCs.: detection of micro-particles
  Interventions: Diagnostic Test: b. Detection of micro particles and their subtypes by flow cytometery on(BECKMAN COULTER CytoFLEX flow cytometer).

INTERVENTIONS:
Diagnostic Test: b. Detection of micro particles and their subtypes by flow cytometery on(BECKMAN COULTER CytoFLEX flow cytometer). — detection of micro-particles

SUMMARY:
Red blood cell (RBC) transfusion is a common therapeutic approach, and almost 85 million packed red blood cells (pRBCs) are transfused annually worldwide.Transfusion efficacy largely depends on the patient's general health, but the composition of transfused pRBCs also can have an impact.

DETAILED DESCRIPTION:
Red blood cell (RBC) transfusion is a common therapeutic approach, and almost 85 million packed red blood cells (pRBCs) are transfused annually worldwide.Transfusion efficacy largely depends on the patient's general health, but the composition of transfused pRBCs also can have an impact. pRBCs are prepared from donated whole blood and can be stored for up to 35 days.During storage, modifications of RBCs occur and affect product quality. Among other changes, these "storage lesions" induce microparticle (MP) formation. MPs are membrane particles measuring 0.1 to 1 µm produced by stimulated or apoptotic cells through modulation of membrane lipid organization and cytoskeleton reorganization. MPs can be produced from any cell type and express antigens characteristic of their original cell. Blood contains platelet-derived MPs (PMPs), which are the most frequent; RBC (erythrocyte)-derived MPs (ERMPs), representing 4% to 8% of total blood MPs; and, more rarely, MPs produced by endothelial cells and leukocyctes. In vivo, aging RBCs release ERMPs over their whole life cycle as a preventive effect of phagocytosis by macrophages. It seems that MPs quickly spread through the body, leading to a variety of biological effects by contact and interactions with many cells. MPs are well-known bioeffectors that mediate strong procoagulant potential, mainly because of phosphatidylserine and tissue factor expression. In this way, MPs are involved in coagulation disorders associated with atherothrombosis and cardiovascular diseases.Their ability to modulate inflammatory and immune responses is increasingly being studied as well as their capacity to carry and transport RNA, DNA, major histocompatibility complex molecules, and infectious agents. Moreover, depending on the type of stimulation that induces MP production, the size and biological functions of the MP can vary.

ELIGIBILITY:
Inclusion Criteria:

* Donors who met criteria of Egyptian National Transfusion Services.
* Serological assays for all blood donors (HBsAgs, HCV antibodies, HIV Ag/Ab and Syphilis antibodies) on Architect i 2000 SR or Centaur XPT (chemoluminescence).

Exclusion Criteria:

* Donors who not met criteria of Egyptian National Transfusion Services.
* Reactive serology.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group 1: 30 filtered backed RBCs. Group 2: 30 non-filtered backed RBCs.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Detection of micro particles and their subtypes by flow cytometery on(BECKMAN COULTER CytoFLEX flow cytometer). - CD235 for red blood cell micro particles. - CD 45 for leukocyte micro particles. - CD41 for platelet micro particles. formation. | 7 days
  Detection of micro particles and their subtypes by flow cytometery on(BECKMAN COULTER CytoFLEX flow cytometer).
  * CD235 for red blood cell micro particles.
  * CD 45 for leukocyte micro particles.
  * CD41 for platelet micro particles.

SECONDARY OUTCOMES:
d. Quantification of micro particles in non filtered packed RBCs (pRBCs) versus filtered (pRBCs) over storage period at 4°C. | 7 days
  Detection of micro particles and their subtypes by flow cytometery on(BECKMAN COULTER CytoFLEX flow cytometer).
  * CD235 for red blood cell micro particles.
  * CD 45 for leukocyte micro particles.
  * CD41 for platelet micro particles.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt